CLINICAL TRIAL: NCT04838067
Title: Validation of Therapeutic Effects of Cefaly on Insomnia by Neuroimaging and Polysomnography Analyses: a Single Site, Single-armed Exploratory Study
Brief Title: Validation of Therapeutic Effects of Cefaly on Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Yoo Hyun Um, Clinical Assistant Professor, Saint Vincent's Hospital, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC18DNSI0145
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefaly Intervention (Experimental): Cefaly
  Interventions: Device: Cefaly

INTERVENTIONS:
Device: Cefaly — Transcutaneous trigeminal nerve electrical neuromodulation

SUMMARY:
The study aims to examine whether the Cefaly has a therapeutic effect on insomnia patients visiting a psychiatric clinic in Korea. The study design is a single site, single-armed exploratory study. Insomnia patients received a 20-minute daily sessions of the Cefaly for 4 weeks. Primary endpoint was a reduction of scores in Pittsburgh Sleep Quality Index, Insomnia Severity Index, Epworth Sleepiness Scale, improvements in polysomnography measures, and changes in resting state networks, cortical thickness, fractional anisotropy and mean diffusivity

DETAILED DESCRIPTION:
Insomnia is well-known for its association with adverse health outcomes. Although insomnia is usually treated with hypnotics or cognitive behavioral therapy for insomnia, the need for novel nonpharmacological treatment for insomnia is increasing emphasized due to reports of side effects and detrimental consequences of hypnotics. Trigeminal nerve electrical neuromodulation has been suggested as a potential treatment modality through its modulation of noradrenergic activity that results in promoting relaxation and reducing hyperarousal. Insomnia patients enrolled in the study will go through a 20-minute daily session of the Cefaly device(originally FDA-approved device for migraine, which electrically modulates trigeminal nerve) for 4 weeks. The objective of this study is to test whether trigeminal nerve electrical neuromodulation has a therapeutic effect, validation measures involving subjective measures(Pittsburgh Sleep Quality Index, Insomnia Severity Index, Epworth Sleepiness Scale), objective measures(Polysomnography measures) and neuroimaging(changes in resting state networks, cortical thickness, fractional anisotropy and mean diffusivity).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have adequately understood the whole study procedures within age range of 19-64 years
2. Patients with insomnia severity index (ISI) score of more than 15

Exclusion Criteria:

1. Cognitive impairment
2. Psychiatric disorders or neurological disorders.
3. Unstable medical conditions
4. Prior diagnosis of sleep disorders
5. Hypnotic prescription
6. History of brain or facial trauma within 3 months
7. Skin abrasions
8. Acrylic acid allergy
9. Electromagnetic hypersensitivity
10. Apnea hypopnea index of >15/hour in the baseline polysomnography.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index(PSQI) | 4 weeks after intervention
  Changes in Pittsburgh sleep quality index scores PSQI global score of more than 5 signifies major sleep disturbance, higher scores suggesting greater sleep disturbance.
Insomnia severity index(ISI) | 4 weeks after intervention
  Changes in Insomnia severity index scores ISI is a brief, self-rated scale that is widely used to measure insomnia severity. With seven items scored on a 0-4 scale, it only takes about 5 minutes to complete and scores of 15 or more indicates insomnia of moderate to severe severity.
Epworth sleepiness scale(ESS) | 4 weeks after intervention
  Changes in Epworth sleepiness scale scores Score of more than 10 signifies clinically meaningful daytime sleepiness, with higher scores indicating more severe sleepiness.
Polysomnography measures-1 (Total sleep time) | 4 weeks after intervention
  Changes in Total sleep time
Polysomnography measures-2 (Wake after sleep onset) | 4 weeks after intervention
  Changes in Wake after sleep onset
Polysomnography measures-3( Stage 1 sleep period) | 4 weeks after intervention
  Changes in Stage 1 sleep period
Polysomnography measures-4(Stage 2 sleep period) | 4 weeks after intervention
  Changes in Stage 2 sleep period
Polysomnography measures-5(Stage 3 sleep period) | 4 weeks after intervention
  Changes in Stage 3 sleep period
Polysomnography measures-6(Total rapid eye movement sleep period) | 4 weeks after intervention
  Changes in Total rapid eye movement sleep period
Polysomnography measures-7(Rapid eye movement sleep latency) | 4 weeks after intervention
  Changes in Rapid eye movement sleep latency
Polysomnography measures-8(Sleep latency) | 4 weeks after intervention
  Changes in Sleep latency
Polysomnography measures-9(Apnea hypopnea index) | 4 weeks after intervention
  Changes in Apnea hypopnea index
Neuroimaging parameter changes-1(Resting state network functional connectivity) | 4 weeks after intervention
  Resting state network functional connectivity changes
Neuroimaging parameter changes-2(Cortical thickness) | 4 weeks after intervention
  Changes in Cortical thickness
Neuroimaging parameter changes-4(Fractional anisotropy) | 4 weeks after intervention
  Changes in Fractional anisotropy
Neuroimaging parameter changes-5(Mean diffusivity) | 4 weeks after intervention
  Changes in Mean diffusivity

CONTACTS AND LOCATIONS:
Overall Officials: Se-Min Choung, Study Director — CMC IRB
Locations (1):
- St.Vincent's Hospital, the Catholic University of Korea, Suwon, South Korea

REFERENCES:
- [Derived] Um YH, Wang SM, Kang DW, Kim NY, Lim HK. Alterations of Resting-State Locus Coeruleus Functional Connectivity After Transdermal Trigeminal Electrical Neuromodulation in Insomnia. Front Psychiatry. 2022 May 10;13:875227. doi: 10.3389/fpsyt.2022.875227. eCollection 2022. PMID 35619611
- [Derived] Um YH, Wang SM, Kang DW, Kim NY, Lim HK. Impact of transdermal trigeminal electrical neuromodulation on subjective and objective sleep parameters in patients with insomnia: a pilot study. Sleep Breath. 2022 Jun;26(2):865-870. doi: 10.1007/s11325-021-02459-0. Epub 2021 Aug 12. PMID 34383274

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT04838067/SAP_000.pdf